CLINICAL TRIAL: NCT01749202
Title: Effects of Stearidonic Acid-Containing Foods on Eicosapentaenoic Acid Levels in Red Blood Cells and Omega-3 Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solae, LLC (Industry)
Collaborators: Provident Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRV-10001
Record Dates: First submitted 2012-06-15; First posted 2012-12-13 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Sudden Cardiac Death; Sudden Cardiac Arrest; Cardiovascular Disease
Keywords: Omega 3 fatty acids; Omega 3 Index; Stearidonic acid (SDA); Red Blood Cells; Lipids
MeSH Terms: conditions — Death, Sudden, Cardiac; Cardiovascular Diseases | interventions — Food

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Negative Control (Placebo Comparator)
  Interventions: Dietary Supplement: Sunflower Oil Softgels; Other: Sunflower Oil Food
- Positive Control (Active Comparator)
  Interventions: Dietary Supplement: EPA softgels; Other: Sunflower Oil Food
- Active (Experimental)
  Interventions: Dietary Supplement: Sunflower Oil Softgels; Other: SDA soybean Oil Food

INTERVENTIONS:
Dietary Supplement: Sunflower Oil Softgels — 3 x 500 mg softgel capsules/day
  Arms: Active; Negative Control
Dietary Supplement: EPA softgels — 3 x 500 mg softgel capsules/day
  Arms: Positive Control
Other: Sunflower Oil Food — 3 servings/day
  Other Names: Food
  Arms: Negative Control; Positive Control
Other: SDA soybean Oil Food — 3 servings/day
  Other Names: Food
  Arms: Active

SUMMARY:
The purpose of this study is to assess the effect of stearidonic acid when used as a food ingredient on eicosapentaenoic enrichment of red blood cell membranes and Omega-3 Index in men and women.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 21 to 65 years of age.
2. BMI) ≥18.00 and <40.00 kg/m2.
3. No health conditions that would prevent him/her from fulfilling the study requirements as judged by the Investigator on the basis of medical history and routine laboratory test results.
4. Willing to avoid alcohol consumption for 24 h prior to every clinic visit.
5. No plans to change smoking habits during the study period.
6. Willing to maintain a stable body weight, activity level and dietary pattern except for use of the study products, as directed.
7. Understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Subject has coronary heart disease or a coronary heart disease risk equivalent including any of the following:

   * Diabetes mellitus
   * Clinical signs of atherosclerosis including peripheral arterial disease, abdominal aortic aneurysm, carotid artery disease
   * Presence of multiple risk factors that give a person a greater than 20% chance for developing coronary artery disease within 10 years.
2. Abnormal laboratory test results of clinical significance
3. TG ≥400 mg/dL at visit 1, week -2.
4. Smokes more than one pack of cigarettes (20 cigarettes) per day.
5. History or presence of clinically important renal, hepatic, pulmonary, biliary, gastrointestinal, neurologic or endocrine disorders that in the judgment of the Investigator, would interfere with the subject's ability to provide informed consent, comply with the study protocol Stable, treated hypothyroidism is allowed.
6. Uncontrolled hypertension
7. Unstable use within four weeks of visit 1 (week -2) of antihypertensive medications or thyroid hormone replacement.
8. Use of any lipid-altering drugs, including statins, bile acid sequestrants, cholesterol absorption inhibitors, fibrates, or prescription formulations of niacin within four weeks of visit 1 (week -2) and throughout the study. If a subject needs to wash off of a drug, he/she will be consented and then asked to return after the four week washout.
9. Use of EPA/DHA from a drug or supplement within four months of visit 1
10. Frequent use (more than twice per month) of any non-study-related EPA/DHA containing enriched foods (such as DHA-enriched eggs) within four months of visit 1, week -2 and avoidance of these enriched foods throughout the study period
11. Use of seeds and oils containing a significant amount of ALA
12. Consumption of fatty fish (salmon, herring, mackerel, albacore tuna, or sardines) more than twice per month
13. Use of any dietary supplement known to alter lipid metabolism
14. Use of any weight-loss medication
15. Use of any weight loss supplement or program within four weeks of visit 1
16. Known allergy or sensitivity to study products or any ingredients of the study products.
17. Subject is unwilling to consume the study products (bars, beverages and capsules) based on results from the taste testing of the study products at visit 1, week -2.
18. Subject has a history or presence of cancer in the prior two years, except for non-melanoma skin cancer
19. Females who are pregnant, planning to be pregnant during the study period, lactating, or women of childbearing potential who are unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation.
20. Current or recent history of (within 12 months of visit 1, week -2) or strong potential for alcohol or substance abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1 ½ oz distilled spirits).
21. Exposure to any non-registered drug product within 30 days prior to the screening visit (visit 1, week -2).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
End of treatment EPA level in RBC membranes, expressed as a percent of total RBC membrane fatty acids | 12 weeks

SECONDARY OUTCOMES:
Omega-3 Index | 12 weeks
SDA percent of total RBC membrane fatty acids | 12 weeks
Triglycerides | 12 weeks
Fasting insulin | 12 weeks
HOMA (IR) and HOMA (%B) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ratna Mukherjea, PhD, Principal Investigator — Solae, LLC
Locations (1):
- Provident Clinical Research &Consulting, Glen Ellyn, Illinois, United States